CLINICAL TRIAL: NCT02090309
Title: The Association Between Low Cortisol Level and Whiplash Syndrome and the Effect of a Single Hydrocortisone Injection on Neck Symptoms Among Motor Vehicle Accident Victims: a Randomized Placebo Controlled Double Blinded Study
Brief Title: Association Between Low Cortisol Levels and Whiplash Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: sor0237-13ctil
Record Dates: First submitted 2014-02-11; First posted 2014-03-18 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-01

CONDITIONS: Injuries, Whiplash
MeSH Terms: conditions — Whiplash Injuries | interventions — Hydrocortisone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydrocortisone injection (Active Comparator): I.V Hydrocortisone 100 mg single bolus.
  Interventions: Drug: Hydrocortisone
- normal saline (Placebo Comparator): I.V normal saline 0.9% a single bolus of 5 ml.
  Interventions: Drug: normal saline 0.9%

INTERVENTIONS:
Drug: Hydrocortisone — 100 mg IV (in the vein) injection as a single bolus of hydrocortisone for the study group.
  Other Names: Cortisol
  Arms: Hydrocortisone injection
Drug: normal saline 0.9% — IV injection of 5 ml normal saline 0.9% as a single bolus.
  Arms: normal saline

SUMMARY:
The investigators hypothesis is that low (or low relatively to the situation) cortisol levels might be a causative factor of whiplash injury or post traumatic stress disorder following road accidents. In this study the investigators enroll patients who sustained a road accident. From all patients a blood sample will be withdrawn to measure cortisol concentrations. Than, the patients will be divided into 2 groups: the study group will receive a single injection of intravenous Hydrocortisone 100 milligram (a synthetic steroid used routinely for many years). The control group will receive a same volume of normal saline which would be used as a placebo treatment. The investigators assume that patients with low cortisol levels would tend to have a higher incidence of whiplash injuries and / or post traumatic stress disorders, and that a single bolus of hydrocortisone may prevent these untoward sequelas of trauma.

DETAILED DESCRIPTION:
Study protocol Patients arriving during day time (08:00 - 16:00) to the Soroka Hospital emergency department following a motor vehicle accident and will be found eligible will be asked to participate in the study. Following an informed consent the recruited patients will be randomly divided into a study group or a control group. From all the participants a volume of 5 milliliter of peripheral blood will be withdrawn for cortisol concentration determination prior to the study intervention. After withdrawing the blood sample patients will receive a single bolus of intravenous Hydrocortisone 100 milligram (study group) or normal saline (0.9%) at a similar volume to that of the study drug, 5 ml (control group). Patients will be otherwise receiving the regular management of a trauma patient. The enrolled patients will fill simple, short questionnaires including demographic data, neck disability index, (NDI), numeric pain rating scale (NPRS), Tampa scale for kinesiophobia (TSK-11), PTSD questionnaire (PDA), and will be assessed by the treating physician for the degree of whiplash (WAD 0-4).

The patients will be followed-up by one of the investigators for a period of 6 months. In each visit the patient will be assessed again by the above mention tools.

Sample size: 45 patients in each arm. Blinding and randomization: triple blinding and using a randomization software. Statistical assessment will be performed to identify differences of developing WAD (whiplash associated disorder) between patients who had an admission low level of cortisol compared with those who had a high or normal level, and also between patients who received hydrocortisone compared to those who received placebo.

ELIGIBILITY:
Inclusion Criteria:

* victims of motor vehicle accidents
* signed informed consent

Exclusion Criteria:

* pregnancy
* traumatic brain injury
* psychiatry disorders
* active cancerous conditions
* adrenal diseases
* medical treatment by estrogens, anti-depressants, melatonin, pain control.
* substance abuse
* hospitalization due to the trauma
* contra indication to hydrocortisone treatment
* over 6 hours from time of injury

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Prevention of whiplash syndrome according to validated scales of pain and neck motion disability. | Six months following the motor vehicle accident.
  Accomplishment of the primary outcome is measured by a composite of several variables. The following indices will be used to measure the primary outcome among the enrolled patients: neck disability index, numeric pain rating scale, Tampa scale for kinesiophobia, PTSD questionnaire (PDA), and will be assessed by the treating physician for the degree of whiplash (0-4).

CONTACTS AND LOCATIONS:
Overall Officials: David Czeiger, M.D. PhD, Principal Investigator — Soroka University Medical Center
Locations (2):
- Israel (2):
  - Soroka Medical Center, Beersheba, Negev
  - Soroka University Medical Center, Beersheba, Negev

REFERENCES:
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for prevention of post-traumatic stress disorder (PTSD) in individuals experiencing acute traumatic stress symptoms. Cochrane Database Syst Rev. 2024 May 20;5(5):CD013613. doi: 10.1002/14651858.CD013613.pub2. PMID 38767196
- [Derived] Bertolini F, Robertson L, Bisson JI, Meader N, Churchill R, Ostuzzi G, Stein DJ, Williams T, Barbui C. Early pharmacological interventions for universal prevention of post-traumatic stress disorder (PTSD). Cochrane Database Syst Rev. 2022 Feb 10;2(2):CD013443. doi: 10.1002/14651858.CD013443.pub2. PMID 35141873
- [Derived] Shaked G, Shaked D, Sebbag G, Czeiger D. The effect of steroid treatment on whiplash associated syndrome: a controlled randomized prospective trial. Eur J Trauma Emerg Surg. 2021 Aug;47(4):1115-1122. doi: 10.1007/s00068-019-01282-3. Epub 2019 Dec 6. PMID 31811333